CLINICAL TRIAL: NCT02800161
Title: Trehalose as add-on Therapy in Bipolar Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Consorcio Centro de Investigación Biomédica en Red (CIBER) (Other Government)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: #14t-012
Record Dates: First submitted 2016-05-09; First posted 2016-06-15 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2021-08

CONDITIONS: Bipolar Disorder; Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — Trehalose; Maltose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trehalose (Active Comparator): Trehalose 70g/die
  Interventions: Drug: Trehalose
- Placebo (Placebo Comparator): Maltose 70g/die
  Interventions: Drug: Maltose

INTERVENTIONS:
Drug: Trehalose — Trehalose 70g/die
  Arms: Trehalose
Drug: Maltose — Maltose 70g/die
  Arms: Placebo

SUMMARY:
The ongoing research on bipolar disorder (BD) has highlighted its pervasive and debilitating nature, characterized by lifelong recurrent episodes and residual intraepisodic symptomatology. Epidemiologic, comorbidity, cost-of illness, and mortality studies have reported dramatic illness-associated morbidity and premature mortality in bipolar patients. The efficacy and safety of antidepressant drug treatment in BD is the subject of long-standing debate based on a scientific literature that is limited and inconsistent. The evidence base for the use of antidepressant drugs in BD is strikingly weak, and there is insufficient evidence for treatment benefits with antidepressants combined with mood stabilizers. The need to develop new agents for the treatment of depression, and in particular bipolar depression, with better efficacy and/or tolerability, remains unmet. In the past years there has been increasing interest in the health benefits of supplemental and/or dietary substances in the treatment and prevention of depression. The disaccharide trehalose protects cells from hypoxic and anoxic injury and suppresses protein aggregation. In vivo studies with trehalose show cellular and behavioural beneficial effects in animal models of neurodegenerative diseases. Moreover, trehalose was shown to enhance autophagy, a process that had been recently suggested to be involved in the therapeutic action of antidepressant and mood-stabilizing drugs. In fact, trehalose may have antidepressant-like properties and that the trehalose induced behavioral changes are possibly related to trehalose effects to enhance autophagy. Furthermore, preliminary data indicates that trehalose also augments lithium effects in animal models (mice). Based on this hypothesis, this project aims to conduct a study to assess the efficacy and tolerability of trehalose as adjunctive treatment to lithium in bipolar depression.

DETAILED DESCRIPTION:
This is an investigator-initiated parallel group pilot study. All patients will give a signed informed consent prior to initiation of any study procedure.

Study setting: This unicentric pilot study will be carried out at the Bipolar Disorder Programme of the Hospital Clinic, University of Barcelona. Over 700 Bipolar Disorder patients are currently treated by Bipolar Disorders Program of the Hospital Clinic and University of Barcelona, a tertiary center providing integrated care for patients from a specific catchment area as well as difficult-to-treat bipolar patients derived from all over Spain, as already described elsewhere.

Patients are considered to be enrolled in the study when they sign the informed consent. Patients are considered to be randomized when they are assigned to receive either trehalose or maltose. It is expected that at least 60 patients will be randomly assigned in a 1:1 ratio of trehalose 70g to placebo (maltose 70g). Patients will receive no economic compensation for their participation in the study.

Patients will be evaluated at baseline and at weeks 2, 4 and 6. At baseline, patients will receive explanations regarding the study; after signing the informed consent patients will be interviewed by the study psychiatrist and will be administered the study scales M.I.N.I. International Neuropsychiatric Interview-Plus (MINI-Plus), Montgomery-Asberg Depression Rating Scale (MADRS), Hamilton Rating scale for Depression (HAMD), Clinical Global Impression-Bipolar Disorder (CGI-BP), World Health Organization-well being (WHO-wb), Functioning Assessment Short Test (FAST), Cognitive complaints in bipolar disorder rating assessment (COBRA). Furthermore, patients will undergo routine blood analysis including glycaemia, thyroid function (T3, T4, TSH) as well as lithaemia, at baseline and at week 6. At weeks 2 and 4 patients will be administered MADRS, HAMD, CGI-BP, WHO-wb and FAST scales, and eventual side effects will be recorded. At week 6, patients will be interviewed and MADRS, HAMD, CGI-BP, and FAST and will be administered and side effects recorded. At the final visit (week 6), patients will undergo a clinical interview, followed by administration of MADRS, CGI-BP, WHO-wb, COBRA and FAST scales. Full blood analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar I and II patients aged between 18 and 65.
* Bipolar disorder type I or II and a current major depressive episode (Montgomery-Asberg Depression Rating Scale (MADRS) ≥18.
* Clinical Global Impression-Bipolar version (CGI-BP)≥4.
* All patients need to be receiving lithium at a steady dose (0.5-1.2 mmol/L) during at least 2 weeks prior to the study.
* Other mood stabilizers added to lithium are permitted but at steady dose during at least 2 weeks prior to the study.
* Other psychopharmacological treatments should be at stable dose 2 weeks prior to the study.

Exclusion Criteria:

* Exclusion criteria will be the presence of psychotic features, severe suicidal ideation (score of ≥5 on item 10 of MADRS).
* A severe personality disorder suggesting noncompliance.
* Diabetes Mellitus, any severe neurologic or other somatic illness and the use of somatic medication that could influence the mood.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2022-10 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
Primary Outcome: efficacy assessed with the Montgomery-Asberg Depression Rating Scale (MADRS) | Mean change from baseline to endpoint (week 8)
  The primary outcome measure is evaluation of efficacy in terms of the mean change from baseline in the total score of the Montgomery-Asberg Depression Rating Scale (MADRS) after the 8 weeks of the study.
Primary Outcome: efficacy assessed with the Hamilton Rating scale for Depression (HAMD) | Mean change from baseline to endpoint (week 8)
  The primary outcome measure is evaluation of efficacy in terms of the mean change from baseline in the total score of the Hamilton Rating scale for Depression (HAMD) after the 8 weeks of the study.

SECONDARY OUTCOMES:
Secondary Outcome: response to treatment defined as a reduction of at least 50% on the MADRS (Montgomery-Asberg Depression Rating Scale). | Mean change from baseline to endpoint (week 8)
  Secondary outcome measures will be response treatment defined as a reduction of at least 50% on the MADRS (Montgomery-Asberg Depression Rating Scale) from baseline to endpoint determination at 8 week.
Secondary Outcome: response to treatment defined as a reduction of at least 50% on the HAMD (Hamilton Rating scale for Depression). | Mean change from baseline to endpoint (week 8)
  Secondary outcome measures will be response treatment defined as a reduction of at least 50% on the HAMD (Hamilton Rating scale for Depression) from baseline to endpoint determination at 8 week.
Secondary Outcome: response to treatment defined as a reduction of at least 50% on the CGI-BP (Clinical Global Impression-Bipolar Disorder). | Mean change from baseline to endpoint (week 8)
  Secondary outcome measures will be response treatment defined as a reduction of at least 50% on the CGI-BP (Clinical Global Impression-Bipolar Disorder) from baseline to endpoint determination at 8 week.

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Vieta, MD,PhD, Principal Investigator — Principal Investigator CIBER
Locations (1):
- Hospital Clinic of Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes